CLINICAL TRIAL: NCT02763930
Title: Study of the Impact of Low Fat Dairy (Milk) and High Fat Dairy (Cheese) Consumption on Daytime Ambulatory Blood Pressure and Other Cardiometabolic Risk Factors
Brief Title: Study of the Impact of Low Fat Dairy and High Fat Dairy Consumption on Daytime Ambulatory Blood Pressure
Acronym: GABA2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Agriculture and Agri-Food Canada (Other Government); Dairy Farmers of Canada (Other)
Responsible Party: Principal Investigator, Benoit Lamarche, Professor, Laval University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: INAF-2015-268
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Hypertension
Keywords: Cardiovascular disease; Blood pressure; Hypertension; Dairy products; Milk; Cheese
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CONTROL (dairy-free) (Experimental): 6 weeks experimental diet with all meals and foods provided to participants. The diet contain 32% of fat, 11% of saturated fat (SFA), 13% of mono-unsaturated fat (MUFA), 8% of polyunsaturated fat (PUFA) and 15% of proteins.
  Interventions: Other: Control diet
- MILK (low fat dairy) (Experimental): 6 weeks experimental diet with all meals and foods provided to participants including 3 servings/day of milk (1% fat) per 2500 kcal. The diet contain 32% of fat, 11% of SFA, 13% of MUFA, 8% of PUFA and 15% of proteins.
  Interventions: Other: Milk diet
- GABA-rich cheese (high-fat dairy ) (Experimental): 6 weeks experimental diet with all meals and foods provided to participants including 50g/day of GABA-rich cheddar cheese (approximately 32% fat). The diet contain 32% of fat, 13% of SFA, 13% of MUFA, 6% of PUFA and 15% of proteins.
  Interventions: Other: GABA-rich cheese diet

INTERVENTIONS:
Other: Control diet
  Arms: CONTROL (dairy-free)
Other: Milk diet
  Arms: MILK (low fat dairy)
Other: GABA-rich cheese diet
  Arms: GABA-rich cheese (high-fat dairy )

SUMMARY:
Market trends depicted by Agriculture and Agri-Food Canada suggest stagnation in cheese consumption, with potentially important impact on this key industry in Canada. This is in part due to the commonly accepted notion that saturated fat in the diet, of which cheese contributes significantly, increases the risk of heart disease. Yet, a rather large body of recent evidence suggests that saturated fat may have been unfairly demonized and that its impact on the risk of heart disease may in fact be less important than originally thought. This concept that dairy fat increases the risk of heart attacks therefore needs to be revisited.

The proposed research is designed to investigate which risk factors for heart disease (e.g. cholesterol, blood pressure) are beneficially modified when low fat (milk) and high fat (cheese) dairy products are consumed.

Our hypotheses are : (1) Consumption of low fat dairy (milk 1% fat) compared with a dairy-free control diet reduces daytime ambulatory systolic blood pressure and reduces inflammation; (2) Consumption of a high fat dairy (GABA-rich cheese) compared with a dairy-free control diet reduces daytime ambulatory systolic blood pressure and has favorable effects on LDL particle size, inflammation and HDL-C concentration.

DETAILED DESCRIPTION:
This is a single-center randomized crossover controlled feeding study. Briefly, adult men and women will be recruited based primarily on blood pressure criteria in the Quebec City metropolitan area through the media (newspaper, radio) and mailing lists (n=60).

Participants will be randomized to 3 experimental diets of 6 weeks each: 1- CONTROL dairy-free diet, 2- low fat dairy (MILK, 1% fat, 3 servings/d), 3- high-fat dairy (GABA-rich cheddar cheese, approximately 32% fat, 1 serving (50g)/d). Usual energy intake will be estimated at the beginning of the study using validated tools. Experimental diets will be provided as part of a full feeding protocol under carefully controlled isocaloric conditions to maintain body weight constant. All meals and foods will be provided to participants so that control for energy and macronutrient intake will be optimized. The breakfast meal will represent approximately 30% of the daily energy intake whereas the lunch and dinner meals each will provide 35% of daily energy intake. Participants will be instructed to consume their entire meals. A seven-day cyclic menu will be used. We have opted to test the impact of dairy intake over a 6-week period (as opposed to 4 or 5 weeks) to maximize the chance to observe clinically meaningful changes in blood pressure. Diets will be separated by a 4 to 8 week washout period. Randomization will be stratified by sex. Blood samples will be collected the day before each dietary phase and on 2 consecutive days after each dietary phase. The mean of the 2 consecutive measurements will be used in the analyses.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age between 18 and 75 years
* Average daytime systolic blood pressure ≥ 125 mmHg (blood pressure medication must be stopped 2 weeks before the start of the study).
* Stable weight for 3 months before the start of the study (+/- 5lbs)

Exclusion Criteria:

* Men or women aged under 18 years or over 75 years
* Average daytime systolic blood pressure ≥ 160 mmHg
* Average daytime diastolic blood pressure ≥ 110 mmHg
* History of cardiovascular disease, type 2 diabetes or dyslipidaemia monogenic
* Endocrine disorders
* Regular smoker
* Lipid lowering medications or diabetes medications
* Food allergies and aversions to any food in the composition of experimental menus
* Subjects with special dietary habits (e.g. vegetarianism)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Variation in daytime ambulatory systolic blood pressure after dairy product consumption (Milk or GABA-rich cheese) compared with the control dairy-free diet. | 6 weeks (end-point value)

SECONDARY OUTCOMES:
Variation in lipid concentrations (LDL-C, HDL-C, TG) | 6 weeks (end-point value)
Variation in apolipoprotein B (ApoB) concentration | 6 weeks (end-point value)
Variation in Low Density Lipoproteins (LDL) particle size | 6 weeks (end-point value)
  Post-diet values will be compared
Variation in High Density Lipoproteins (HDL) particle size | 6 weeks (end-point value)
Variation in C-Reactive Protein (CRP) concentration | 6 weeks (end-point value)
Variation in Adiponectin concentration | 6 weeks (end-point value)

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Lamarche, PhD, Principal Investigator — Laval University
Locations (1):
- Institute of Nutrition and Fonctional Foods, Québec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rancourt-Bouchard M, Gigleux I, Guay V, Charest A, Saint-Gelais D, Vuillemard JC, Lamarche B, Couture P. Effects of regular-fat and low-fat dairy consumption on daytime ambulatory blood pressure and other cardiometabolic risk factors: a randomized controlled feeding trial. Am J Clin Nutr. 2020 Jan 1;111(1):42-51. doi: 10.1093/ajcn/nqz251. PMID 31584063